CLINICAL TRIAL: NCT04845438
Title: Evaluation of Biliary Reflux After Mini-gastric Bypass With Using the Biliary Reflux Index
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Private Healthcare Institution Clinical Hospital RGD-Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: CCH-RR-2020-mo-2
Record Dates: First submitted 2021-04-10; First posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Ulcer, Gastric; Bile Reflux
MeSH Terms: conditions — Stomach Ulcer; Bile Reflux

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hand-sewn gastroenteroanastomosis (Active Comparator)
  Interventions: Diagnostic Test: fibrogastroscopy, biopsy of the gastric mucosa, microscopy biopsy materials, using Bile Reflux Index
- stapler gastroenteroanastomosis (Active Comparator)
  Interventions: Diagnostic Test: fibrogastroscopy, biopsy of the gastric mucosa, microscopy biopsy materials, using Bile Reflux Index

INTERVENTIONS:
Diagnostic Test: fibrogastroscopy, biopsy of the gastric mucosa, microscopy biopsy materials, using Bile Reflux Index — fibrogastroscopy, biopsy of the gastric mucosa, microscopy biopsy materials, using Bile Reflux Index

SUMMARY:
MGB is considered to be the best alternative to Roux-en-Y gastric bypass (RYGB) due to the shorter operation time and fewer possible complications.

The purpose of this study was to determine biliary reflux in patients undergoing MGB/OAGB with a hand-sewn gastroenteroanastomosis, and MGB/OAGB with a stapler gastroenteroanastomosis.

ELIGIBILITY:
Inclusion Criteria:

* morbid obesity
* BMI above 35 kg/m2 with obesity related comorbidity
* BMI above 40 kg/m2
* undergoing MGB/OAGB
* no bile reflux during preoperative period

Exclusion Criteria:

* revisional operations
* therapy-resistant bile reflux during preoperative period
* history of bariatric surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Estimated)
Dates: Start 2020-12-29 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-03-08 (Estimated)

PRIMARY OUTCOMES:
Success | 12 month
  Determination of the BRI index in patients undergoing MGB/OAGB can be used as a screening method for diagnosing biliary reflux in order to prevent and develop tactic for further management of patients from a risk group of complications associated with the toxic effects of an aggressive bile

CONTACTS AND LOCATIONS:
Locations (1):
- Private Healthcare Institution Clinical Hospital "RGD-Medicine" Rostov-on-Don", Rostov-on-Don, Russia

IPD SHARING:
Plan to Share IPD: No